

### STATISTICAL ANALYSIS PLAN

A Multicenter, Prospective, Active Controlled, Real World, Phase 4 Study of EXPAREL® in Multimodal Regimens Compared with Standard of Care for Postsurgical Pain Management in Subjects Undergoing Lumbar Posterior Spine Surgeries (FUSION)

**Protocol No.:** 402-C-413

IND No.: Not applicable

Study Phase: 4

Study Drug: EXPAREL® (bupivacaine liposome injectable

suspension)

**Date/Version:** 19 October 2020/Version 1.0

Prepared by: Ashley Pajak, MS

Pacrira Pharmaceuticals, Inc.

**Sponsor:** Pacira Pharmaceuticals, Inc.

5 Sylvan Way

Parsippany, NJ 07054 Tel: 973-254-3560

### **Confidentiality Statement**

The information contained in this document is confidential and the property of Pacira Pharmaceuticals, Inc. It should not be reproduced, revealed, or sent to third parties other than Institutional Review Boards/Independent Ethics Committees and the Investigator's research support staff participating in the conduct of the study without the prior written authorization of Pacira Pharmaceuticals, Inc.

### **SIGNATURE PAGE**

| | DocuSigned by: | |
|---|---|---|
| | Don Manning | 21-Oct-2020 |
| Approved by: | Signer Name: Don Manging Donald Martenson: Papprove this document Chief Moglinal Office, 201 mice h Operations | Date |
| | E092D856DC394A9B80AB96BC2794DF0F DocuSigned by: | |
| | Michael Rozycki | 19-Oct-2020 |
| Approved by: | Michael Name. Michael Rozycki Michael Rozyckin. Paprove this document Vice Brosing on the Rozyclatron Affairs 1 AM PDT | Date |
| | B4308C39715A4ED49144E886EF300CA3 | |
| | DocuSigned by: | |
| | Gary Mexins | 20-oct-2020 |
| Approved by: | Signer Name: Gary Nevins Gary Signifig Reason: I approve this document Execution Modical Distance Leading Comment | Date |
| | 558D44F13780486C86D569374F58CB46 DocuSigned by: | |
| | Vincent Yu | 19-oct-2020 |
| Approved by: | Signer Name: Vincent Yu | Date |
| ripproved by. | Vince <b>និច្ឆាក់ល្អ Repo</b> n: I approve this document<br>Vice ទ <del>ាំចនាលាក្រាស់ លេខស</del> េស្តិទា l 12:16:02 PM PDT | Dave |
| | 381A73A2808A488ABDBCE0932644F2EC | |

### TABLE OF CONTENTS

| 1. | INTR | ODUCTION | 6 |
|---|---|---|---|
| 2. | STUI | DY OBJECTIVES | 7 |
| | 2.1 | Primary Objective | 7 |
| | 2.2 | Secondary Objectives | 7 |
| 3. | STUI | DY OVERVIEW | 8 |
| 4. | DEFI | NITIONS | 9 |
| 5. | ANA | LYSIS SETS | 9 |
| 6. | STA | FISTICAL METHODS | 10 |
| | 6.1 | General Principles | 10 |
| | | 6.1.1 Handling Missing Values | 10 |
| | | 6.1.1.1 Exposure, Surgery, and Rescue Opioid Medication Date or Time | 10 |
| | 6.2 | Subject Disposition | 10 |
| | 6.3 | Description of Demographics and Baseline Characteristics | 11 |
| | | 6.3.1 Demographics | 11 |
| | | 6.3.2 Baseline Characteristics | 11 |
| | 6.4 | Surgery Characteristics and Prior Staged Procedure | 11 |
| | 6.5 | Intraoperative, Prior, Concomitant, and Other Mediciations | 11 |
| | 6.6 | Medicial History | 12 |
| | 6.7 | Measurements of Treatment Compliance | 12 |
| | 6.8 | Study Drug Exposure | 12 |
| | 6.9 | Efficacy Analysis | 12 |
| | 6.10 | Health Outcomes Assessments | 12 |
| | 6.11 | Safety Analyses | 12 |
| | | 6.11.1 Adverse Events | 12 |
| | 6.12 | Interim Analysis | 13 |
| 7. | SAM | PLE SIZE REVIEW | 14 |
| 8. | REFI | ERENCES | 15 |
| 9. | TIMI | E AND EVENTS SCHEDULE OF STUDY PROCEDURES | 16 |
| | 9.1 | Part 1 | 16 |
| | 9.2 | Part 2- After PACU Arrival | 17 |
| 10. | LAY | OUT OF LISTINGS | 18 |
| 11. | TAB | LE OF CONTENTS FOR LISTING MOCK-UPS | 19 |

### LIST OF ABBREVIATIONS

| Abbreviation | Description |
|--------------|------------------------------------------------|
| ADL | Activities of daily living |
| AE | Adverse event |
| AICC | Corrected Akaike information criterion |
| ASA | American Society of Anesthesiology |
| ATC | Anatomical therapeutic class |
| AUC | Area under the curve |
| BIC | Schwarz's Bayesian information criterion |
| BLOQ | Below the limit of quantification |
| BMI | Body mass index |
| BPI-sf | Brief Pain Inventory – short form |
| bpm | Beats per minute |
| CAS | Color Analog Scale |
| CI | Confidence interval |
| CMP | Complete metabolic panel |
| CRF | Case report form |
| CSR | Clinical study report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CV | Coefficient of variation |
| EMA | European Medicines Agency |
| ER | Emergency room |
| GM | Geometric mean |
| HADS | Hospital Anxiety and Depression Scale |
| HCl | Hydrochloride |
| hr, h | Hour |
| ICF | Informed consent form |
| ICH | International Council for Harmonisation |
| IM | Intramuscular |
| IV | Intravenous |
| LIA | Local infiltration analgesia |
| LOS | Length of stay |
| MCID | Minimum clinically important difference |
| MedDRA | Medical dictionary for regulatory affairs |
| min | Minutes |

| Abbreviation | Description |
|--------------|---------------------------------------------------|
| mg MED | Morphine equivalent dose in mg |
| mg | Milligram |
| MPADSS | Modified Post-Anesthesia Discharge Scoring System |
| n | Number of subjects |
| NCI | National Cancer Institute |
| NRS | Numerical Rating Scale |
| OCC | 5-item Opioid Compliance Checklist |
| ORAE | Opioid-related adverse events |
| OR-SDS | Opioid Related-Symptoms Distress Scale |
| PACU | Post-Anesthesia Care Unit |
| PO | Oral |
| PT | Preferred Term |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SC | Subcutaneous |
| SD | Standard deviation |
| SOC | Standard of care |
| SOPA | Survey of Pain Attitudes |
| TEAE | Treatment-emergent adverse event |
| TLF | Tables, listings and figures |
| USFDA | United States Food and Drug Administration |
| WHO | World Health Organization |
| WHO-DD | World Health Organization – Drug Dictionary |

### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) describes the planned statistical analysis and reporting of the clinical study 402-C-413 titled "A Multicenter, Prospective, Active Controlled, Real World, Phase 4 Study of EXPAREL® in Multimodal Regimens Compared with Standard of Care for Postsurgical Pain Management in Subjects Undergoing Lumbar Posterior Spine Surgeries (FUSION)". This study is intended to evaluate postsurgical opioid consumption in adult subjects receiving EXPAREL and undergoing posterior lumbar spine surgeries.

This study was prematurely terminated by the sponsor. At the time of termination, the study has enrolled 65 subjects.

The purpose of this SAP is to outline how the collected data will be summarized and presented for the abbreviated study report.

The following documents were reviewed in preparation of this SAP:

- Amendment 1 of Protocol 402-C-413 issued on 25 February 2019.
- Case Report Form (CRF) final version 4.0 issued on 06 July 2020.
- ICH Guidance on Statistical Principles for Clinical Trials (E9)

The reader of this SAP is encouraged to also read the clinical protocol and other identified documents for details on the planned conduct of this study. Operational aspects related to the collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analyses.

### 2. STUDY OBJECTIVES

### 2.1 Primary Objective

The primary objective of this study is to compare postsurgical opioid consumption through 72 hours postsurgery in patients receiving local infiltration analgesia (LIA) with EXPAREL and bupivacaine hydrochloride (HCl; EXPAREL group) with that of patients receiving standard of care (SOC; Control group) in adult subjects undergoing posterior lumbar spine surgeries where both groups are receiving a multimodal pain regimen.

### 2.2 Secondary Objectives

The secondary objectives are to:

- 1. Compare safety and effectiveness outcomes following LIA with EXPAREL and bupivacaine HCl versus SOC in adult subjects undergoing posterior lumbar spine surgeries through 72 hours, including time to first opioid, opioid-related adverse events (ORAEs).
- 2. Compare health outcomes following LIA with EXPAREL and bupivacaine HCl versus SOC in adult subjects undergoing posterior lumbar spine surgeries, including discharge readiness, hospital (or other facility) length of stay (LOS), discharge disposition, hospital readmissions, and health service utilization.

### 3. STUDY OVERVIEW

This is a Phase 4, multicenter, prospective, active-controlled, real-world study in approximately 225 adult subjects undergoing posterior lumbar spine surgeries under general anesthesia. This will be an open-label study and neither subjects nor investigators will be blinded for study group allocation. This study will include three cohort groups: cohort 1 – open lumbar spinal fusion technique ("open" cohort); cohort 2 – minimally invasive tubular and/or percutaneous pedicle screw insertion for lumbar decompression with or without fusion ("tubular/percutaneous without midline incision" cohort); and cohort 3 – lumbar decompression surgery (LDS) without fusion (discectomy or laminectomy cohort) outpatient cohort.

The initial sample size in each study cohort (i.e., cohort 1, cohort 2 and cohort 3) is estimated at 75 subjects (50 subjects with EXPAREL and 25 subjects with Control group), for a total of 225 subjects in all three cohorts. Within each assigned cohort, subjects will be allocated in a 2:1 ratio to the EXPAREL (50 subjects) and Control group (25 subjects).

The following sequence will be carried out for all cohorts: First, the subjects who meet eligibility criteria will be treated according to the institution's SOC. Their data will be collected prospectively. Next, at each investigational center, the administration of EXPAREL and bupivacaine HCl to the first 1 to 3 subjects in each cohort will be observed to ensure that the correct procedure for infiltration as described in the infiltration guide is being followed. If the infiltration was performed correctly, the subject will be included in the study. If the infiltration was performed incorrectly, the subject will continue in the study but will be removed from statistical analysis and will be replaced to ensure at least 50 evaluable EXPAREL patients are enrolled per cohort. If subjects are discontinued for other reasons, they will be replaced such that a total sample size of 75 fully evaluable subjects is obtained in each study cohort, with 50 in the EXPAREL group and 25 in the Control group. Criteria for being fully evaluable will be defined in detail in Section 5.

Figure 1 Study Schema



Source: Protocol, Amendment 1, 25 February 2019

### 4. **DEFINITIONS**

### **Study Day**

Study Day is calculated as the date of the event minus the date of the start of surgery plus one (1), if the date of event is on or after the date of the start of surgery. If the date of the event is before the date of the start of surgery, study day is the date of the event minus the date of the start of surgery.

### Time 0 (zero)

Time 0 is defined as the date and time of the end of surgery.

### **Treatment-emergent Adverse Events**

Treatment-emergent adverse events (TEAEs) are those with onset between the end date and time of surgery, and the end of the study (Study Day 30 or until termination from the study).

### **Baseline**

Baseline measurement or assessment is defined as the last available non-missing measurement or assessment prior to the start of surgery.

### 5. ANALYSIS SETS

All Subjects: all the listings presented in this SAP will be based on all enrolled subjects. Includes the following subjects who enrolled but did not undergo surgery; 101-01-0013, 101-03-0034, 109-02-0001, 113-03-0039.

### 6. STATISTICAL METHODS

### 6.1 General Principles

Only listings of subject data collected during the study will be provided. All listings will be sorted by treatment group, site ID, subject ID, and, if applicable, collection date and time.

### **6.1.1 Handling Missing Values**

Data will be included in the listing as is. No imputed values will be included in the listings. However, in order to provide the drug safety profile, the missing or partial date/time will be imputed only for the determination of treatment emergency or prior/concomitant status.

### 6.1.1.1 Exposure, Surgery, and Rescue Opioid Medication Date or Time

It is expected that all necessary information on study drug exposure and surgery (dates and times) will be complete. Any such information that is missing and cannot be obtained through query resolution may be imputed, on a case-by-case basis, in a conservative manner that minimizes bias.

### 6.1.1.2 Adverse Event or Concomitant Medications Dates or Time.

For adverse events (AEs) or concomitant medications with missing or partially missing start/stop date/time, the following imputation rules will be applied:

For partial start date/time:

- If the year is unknown, then the date will be assigned the year of the start of surgery.
- If the month is unknown, then:
  - o If the year matches the year of start of surgery, then the month and day of the dose of study drug date will be used to impute the missing month and corresponding day.
  - Otherwise, 'January' will be assigned.
- If the day is unknown, then:
  - o If the month and year match the month and year of the dose of start of surgery, then the day of the start of surgery date will be imputed.
  - o Otherwise, '01' will be assigned.
- If the time is unknown, then:
  - o If the date (day, month, and year) matches the date of the start of surgery, then the end time of the surgery will be imputed.
  - Otherwise, '00:00' will be assigned.

For partial stop date/time:

- If the year is unknown, then the date will be assigned the year that subject had surgery, and time will be set to the last time of the day ('23:59').
- If the month is unknown, then month of start of surgery will be assigned.
- If the day is unknown, then the last day of the month will be assigned.
- If the time is unknown, then the last time of the day will be assigned ('23:59'), with the exception of end times for epoch in any CDISC dataset, where next day and '00:00' would be assigned.

### **6.2 Subject Disposition**

A listing of subject disposition will be provided, which will include information on study completion status among others.

### 6.3 Description of Demographics and Baseline Characteristics

### 6.3.1 Demographics

Listing of demographic data will include:

- Initals
- Date of Birth (DOB)
- Age (years)
- Sex
- Ethnicity
- Race

### **6.3.2** Baseline Characteristics

Listing of baseline characteristic data will include:

- Screening Survey of Pain Attitudes (Single-item SOPA)
- Screening Hospital Anxiety and Depression Scale (HADS)
- Screening 5-item Opioid Compliance Checklist (OCC)
- Height (cm)
- Weight (kg)
- Body mass index (BMI;kg/m²)

The formula for BMI is  $w/(h^2)$ , where w is weight in kilograms and h is height in meters. Weight in pounds will be converted to kilograms using the conversion factor of 2.2046 pounds to 1 kilogram. Height in inches will be converted to meters using the conversion factor of 0.0254 meters to 1 inch.

### 6.4 Surgery Characteristics and Prior Staged Procedure

Surgery characteristics include duration of surgery, total incision length, and type of procedure. Duration of surgery is calculated as the difference between the end of surgery and start of surgery times and reported in hours. Surgical characteristics will be included in data listings.

Prior staged procedue characteristics will be included in data listings.

### 6.5 Intraoperative, Prior, Concomitant, and Other Mediciations

Intraoperative, prior, and concomitant medications will be coded using the World Health Organization Drug Dictionary (WHODrug version: march 2019 B3) and will be classified according to the default anatomical therapeutic chemical (ATC 4) classification term and preferred term (PT).

Intraoperative medications are defined as medications given as part of the surgical procedure. These may include anesthesia, opioids or other medications and are collected on the intraoperative medication page of the case report form.

Prior medications are defined as medications with a stop date and time prior to the start of surgery and reported on the prior/concomitant medication page of the case report form.

Concomitant medications are defined as medications taken after the start of surgery (i.e., started prior to the start of surgery and continued after or started after the start of surgery) and reported on the prior/concomitant medication page of the case report form.

Data listings will be created for all medications, with separate listings for intraoperative, prior, concomitant, multimodal pain pre-operative, multimodal pain post-operative, prescription daily pain, and rescue medications.

A listing mapping the ATC class and PT to verbatim term will be presented.

### **6.6 Medicial History**

Relevant medicial history and surgery will be presented in a by-subject listing.

### 6.7 Measurements of Treatment Compliance

Study treatment is administered by a party other than the subject, therefore compliance is assured.

### 6.8 Study Drug Exposure

A listing of study drug exposure, which includes volume of injection administered will be provided.

### **6.9 Efficacy Analysis**

Listing of the following efficacy assessments will be provided:

- Pain intensity score using the NRS
- OR-SDS at 24, 48, and 72 hours postsurgery, at discharge, and at 14 days
- Brief Pain Inventory Short Form at screening/baseline, 24 hours, 48 hours, and 72 hours, at discharge, and at 14 days

### **6.10 Health Outcomes Assessments**

Listing of the following health outcome assessments will be provided:

- Post-Anesthesia Care Unit (PACU)- The date and time of admission and discharge, and the hours spent in the PACU will be provided in a listing. The hours spent in PACU will be computed as the date and time of discharge from PACU minus the date and time of admission to PACU.
- Surgical Facility- The date and time of admission and discharge, and the hours spent in the step-down and surgical facility will be provided in a listing.
- Modified Post-Anesthesia Discharge Scoring System (MPADSS) at 24, 48, and 72 hours, or at discharge, or until the subject attains a score of 9, whichever occurs first.
- Discharge Disposition
- Day 14 Call to doctor and office visits related to pain
- Day 30 Call to doctor and ER visits related to pain, and pain-related/all-casue 30-day readmissions

### **6.11 Safety Analyses**

Safety assessments in this study consist of AEs. Adverse events will be collected from the time of informed consent through to the final Day 30 visit.

### **6.11.1** Adverse Events

All AEs will be mapped to PTs and related system/organ class using the Medical Dictionary for Regulatory Activities (MedDRA Version 22.0).

An AE will be considered TEAE if the onset date and time is between the end time and date of surgery and the final Day 30 visit. An AE will be considered related to study drug if "Possible", "Probable" and "Definite.

If an AE has a partial onset date and time the imputed start and stop dates and times will be used to determine treatment-emergence (e.g., stop date and time is before start time of surgery). If an AE has a missing relationship it will be assumed to be "Related".

A listing of all AEs will be provided, with a flag indicating TEAEs.

### **6.12 Interim Analysis**

Interim analysis may be conducted to adjust to variability. Adaptive study design (i.e., adjustment of sample size, cohort sequence, type of surgical procedure, endpints, etc.) will be used.

### 7. SAMPLE SIZE REVIEW

The sample size for this study was based on the primary outcome measure of postsurgical opioid use in mg MED PO from the end of surgery (closure of wound/incision) until 72 hours postsurgery. Based on preliminary data, the coefficient of variation (CV) is approximately 60%. The minimum clinically important difference (MCID) for this outcome was estimated at 40%.

With these parameters and a beta of 0.2 (i.e., 80% power), an alpha of 0.05, a 2-sided test, and allocating subjects in a 2:1 ratio to the EXPAREL group or Control group to minimize barriers to enrollment for an approved and marketed medication, a total sample size of 75 fully evaluable subjects is required in each study cohort, with 50 subjects in the EXPAREL group and 25 subjects in the Control group. The same assumptions are made across all cohorts. Subjects who undergo the planned surgery and whose infiltration is performed correctly and who are not discontinued early from the study for any other reasons will be fully evaluable. Not fully evaluable subjects should be replaced. Given that this study will have a case observation period for the first few subjects in EXPAREL group, if observation is deemed correct and infiltration was performed correctly, subject can be included in the study. If observation is deemed incorrect and infiltration was performed incorrectly, subject will continue in the study but will be removed from statistical analysis and will be replaced to ensure at least 50 evaluable EXPAREL arm patients are enrolled per cohort. The total number of subjects in all three cohorts will be 225, with 150 in the EXPAREL group and 75 in the Control group. This is subject to adjustment per interim analysis if necessary.

### 8. REFERENCES

- 1. American Statistical Association. Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, 07 August 1999. http://www.amstat.org/profession/ethicalstatistics.html
- 2. Rubin, DB. (1987). Multiple Imputation for Nonresponse in Surveys. New York: John Wiley & Sons.
- 3. US Federal Register. International Conference on Harmonisation; Guidance on Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration [Docket No. 97D-0174]. Federal Register Volume 63, Number 179, pages 49583-49598. 16 September 1998.
- 4. Royal Statistical Society. The Royal Statistical Society: Code of Conduct, August 1993. http://www.rss.org.uk/about/conduct.html.

# 9. TIME AND EVENTS SCHEDULE OF STUDY PROCEDURES

### 9.1 Part 1

| Study Procedure | Screening/Baseline<br>(1-30 days prior to surgery) | Pre-op | Тпітя-ор | PACU | Post-op |
|---|---|---|---|---|---|
| Screening and Baseline | | | | | |
| Obtain signed ICF* | × | | | | |
| Record medical and surgical history | × | | | | |
| Record medication history <sup>b</sup> | × | | | | |
| Record demographics and baseline characteristics | × | | | | |
| Record opioid use in last 30 days to determine mg MED PO/day average | x | | | | |
| Record height, weight, and BMI | × | | | | |
| Confirm eligibility | × | | | | |
| Unne pregnancy test (UPT) (for women of childbearing potential) | × | | | | |
| NRS for pain at the pre-surgical area | × | | | | |
| Survey of Pain Attitudes (Single-item SOPA) | x | | | | |
| Brief Pain Inventory – short form (BPI-sf) | × | | | | |
| Hospital Anxiety and Depression Scale (HADS) | × | | | | |
| 5-item Opioid Compliance Checklist (OCC) <sup>e</sup> | × | | | | |
| Record AEs and medications to treat AEs from the time ICF was signed | • | | | | † |
| Day of surgery | | | | | |
| Confirm eligibility; UPT does not need to be repeated | | X | | | |
| Administer scheduled presurgical medications | | X | | | |
| Record surgery start and stop times | | | X | | |
| Prepare study drug | | | X | | |
| Administer study drug, record start and stop times | | | х | | |
| Record intraoperative opioids administered and doses, and all concomitant medications | | | X | | |
| Record times and doses of all opioid and non-opioid rescue medications administered | | | X | | |
| Post-surgery <sup>d</sup> | | | | | |
| Record date, time, and dose of rescue postsurgical analgesics | | | | | X |
| Record date, times, and doses of all multimodal scheduled medications administered | | | | | X |
| Record date, time of admission to, and time of discharge from different hospital units (PACU step-down) | | | | Х | |
| Racond concernitant madications | | ļ | | | 1 |
| Mecong concomitant meatcanons | | , | | | |

Abbreviations: AE = Adverse event; BMI = Body mass index; BPI-sf = Brief Pain Inventory - short form; HADS = Hospital Anxiety and Depression Scale; ICF = Informed consent form; MED = Morphine equivalent dosing; OCC = 5-item Opioid Compliance Checklist (Jamison 2014; Jamison 2016); PACU = Post-anesthesia care unit; PO = per os (oral); SOC = standard of care; SOPA = Survey of Pain Attitude; UPT = urine pregnancy test.

conduct of any screening procedures that are not considered SOC at the institution and such procedures may not be performed until written informed consent is provided. All screening procedures that are not SOC must be performed and documented within the 30-day time window (inclusive of the day of surgery for those subjects who can only be screened on the day of surgery) as described here. During the screening visit, subjects will be assessed for any past or present medical conditions that in the opinion of the investigator would \*No more than 30 days should pass between signing of the ICF and performance of the surgery. Subjects will be screened within 30 days prior to surgery, screening on the day of surgery will be allowed but is discouraged. If a subject can only be screened on the day of surgery, the informed consent process must still be started at least 24 hours prior to the preclude them from study participation.

Record any medications for the condition for which the procedure is being performed that were administered within 30 days prior to screening.

<sup>6</sup> Sources for 5-item OCC are Jamison 2014 and Jamison 2016.

All assessments conducted after baseline (prior to the study drug administration) will be timed from the end of surgery. Postsurgical is defined as a period after the end of surgery. End of surgery is defined as the time (when the last incision/wound is closed).

## 9.2 Part 2- After PACU Arrival

| | | | | Ē | rom End<br>6-72 I | From End of Surgery<br>6-72 Hours* | Ţ. | | | Phone Discharge call or Visit* | Phone<br>call or<br>Visit* | Phone<br>call <sup>b</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point 6 hrs ± Time window ±1 hr | 6 hrs<br>±1 hr | 12 hrs<br>±1 hr | | 24 hrs<br>±1 hr | 24 hrs 30 hrs<br>±1 hr ±2 hr | 18 hrs 24 hrs 30 hrs 36 hrs 42 hrs 48 hrs 72 hrs<br>±1 hr ±1 hr ±2 hr ±2 hr ±2 hr ±4 hr <sup>3</sup> | 42 hrs<br>±2 hr | 48 hrs 72 hrs<br>±2 hr ±4 hr <sup>b</sup> | 72 hrs<br>±4 hr <sup>b</sup> | | 14 days 30 days<br>±3 days ±3 days | 14 days 30 days<br>±3 days ±3 days |
| Study Procedure | | | | | | | | | | | | |
| NRS for pain at surgical site | Х | Х | Х | X | Х | Х | Х | Х | Х | Х | X | |
| BPI-sf | | | | × | | | | × | × | × | × | |
| Record date and time of all opioid and non-opioid rescue | | | | | | | | | | | 4 | |
| medications* | | | | | | | | | | | 1 | |
| OR-SDS | | | | X | | | | Х | Х | Х | X | |
| MPADSS* | | | | X | | | | X | X | $X_c$ | | |
| Record date and time of discharge | | | | | | | | | | × | | |
| Record subject discharge disposition | | | | | | | | | | X | | |
| Document any unscheduled phone calls or office visits related to | | | | | | | | | | | | |
| pain | | | | | | | | | | | X | |
| Document any requests for refills for opioid medication | | | | | | | | | | | X | |
| Record persistent opioid use by asking the subject "Are you | | | | | | | | | | | | |
| currently taking opioid medication to manage pain from your | | | | | | | | | | | | |
| spine surgery?" | | | | | | | | | | | | × |
| Document any hospital readmissions related to pain | | | | | | | | | | | | X |
| Document hospital readmissions for any cause | | | | | | | | | | | | X |
| Document any unscheduled visits to the ER related to pain | | | | | | | | | | | | Х |
| Record date and time of AEs and medications to treat AEs | • | | | | | | | | | | | 1 |
| (with dosage) | , | | | | | | | | | | | 1 |

Abbreviations: AE=adverse event; BPI-sf = Brief Pain Inventory - short form; ER = Emergency room; hr/hrs = hour(s); MPADSS = Modified Post-Anesthesia Discharge Scoring System; NRS=numeric rating scale; OR-SDS = Opioid-Related Symptom Distress Scale.

complete the 72 hour assessments as EoS assessments. If early termination occurs after discharge but prior to Day 14, Day 14 assessments are to be completed as EoS assessments. Note: Early Termination: Whenever possible, subjects discontinuing the study should complete end of study (EoS) assessments. Subjects discontinuing prior to 72 hours are to If early termination occurs after Day 14 but prior to Day 30, Day 30 assessments are to be completed as EoS assessments.

Every day from discharge through Day 14, subjects are to record in the eDiary any pain medication (date, time, and dose) taken in the prior 24 hours in addition to recording questionnaire responses. Subjects who were lent an eDiary will have to return to the site at 14 days at which time they are to return the device. Subjects who Subjects are to record their responses to subject questionnaires on an electronic device (eDiary) at screening, while in the hospital (or other facility), and at Day 14. used their own device will have a follow-up phone call at Day 14. All subjects will have a follow up call at 30 days after the surgery.

For all subjects, if discharge occurs prior to 72 hours postsurgery, all Discharge assessments are to be performed at the time of discharge. After discharge, all scheduled assessments should be performed at the scheduled time points (i.e., NRS pain assessments at 6, 12, 18, 24, 30, 36, 42, 48, and 72 hours postsurgery; BPI-sf and OR. SDS at 24, 48, and 72 hours; and date, time, and dose of all opioid and non-opioid rescue medications) and recorded in the eDiary.

Discharge readiness via the MPADSS will be assessed at 24, 48, and 72 hours and/or discharge or until the subject attains a score of 9, whichever occurs first.

### 10. LAYOUT OF LISTINGS

Listings will have 10-point font size. The listing will have Times New Roman, Courier New, or SAS Monospace type face. All final listings will be provided in both PDF and Word (or RTF) file formats.

Titles on the Listings should appear as following:

```
Listing 16.2-1.1.1

Subject Disposition- All Subjects

Cohort: Cohort 1; Treatment: EXPAREL
```

The text "Cohort: Cohort 1; Treatment: EXPAREL" refers to the cohort and treatment group. There should be a page break between the cohort and treatment group and should be presented in the order of:

```
Cohort: Cohort 1; Treatment: SOC
Cohort: Cohort 1; Treatment: EXPAREL
Cohort: Cohort 1; Treatment: NOT TREATED
Cohort: Cohort 2; Treatment: SOC
Cohort: Cohort 2; Treatment: EXPAREL
Cohort: Cohort 2; Treatment: NOT TREATED
Cohort: Cohort 3; Treatment: SOC
Cohort: Cohort 3; Treatment: EXPAREL
Cohort: Cohort 3; Treatment: EXPAREL
Cohort: Cohort 3; Treatment: NOT TREATED
```

Listings should be generally ordered by Cohort, Treatment, Site, Subject and Date where applicable. If data is missing in a column, the column may be populated with "-" for reading ease.

### 11. TABLE OF CONTENTS FOR LISTING MOCK-UPS

| Listing 16.2-1.1: Subject Disposition— All Subjects | 21 |
|---|---|
| Listing 16.2-2: Enrollment– All Subjects | 22 |
| Listing 16.2-3: Inclusion/ Exclusion Criteria- Failures Subjects | 23 |
| Cohort: -; Treatment: SCREEN FAILURES | 23 |
| Listing 16.2-4.1: Demographics – All Subjects | 24 |
| Listing 16.2-4.2: Demographics – Screen Failures | 25 |
| Listing 16.2-4.3: Demographics – Subject Enrolled but No Surgery | 26 |
| Listing 16.2-5.1: Baseline Characteristics (Survey of Pain Attitudes (SOPA))– All Subjects | |
| Listing 16.2-5.2: Baseline Characteristics (Hospital Anxiety and Depression Score (HADS))– All | |
| Subjects | |
| Listing 16.2-5.3: Baseline Characteristics (5-Item Opioid Compliance Checklist (OCC) – All Subjects | |
| Listing 16.2-6.1: Pregnancy test- All Female Subects | |
| Listing 16.2-6.2: Pregnancy test- Female Screen Fails | |
| Listing 16.2-7.1: Admission and Discharge- Post-Anesthesia Care Unit (PACU) – All Subjects | |
| Listing 16.2-7.2: Admission and Discharge – Surgical Facility – All Subjects | 33 |
| Listing 16.2-8.1: Surgery Characteristics- Procedure – All Subjects | |
| Listing 16.2-8.2: Surgery Characteristics- Anesthesia- All Subjects | 35 |
| Listing 16.2-8.3: Surgery Characteristics- Autograft– All Subjects | 36 |
| Listing 16.2-8.4: Surgery Characteristics-Prior Staged Procedure – All Subjects | 37 |
| Listing 16.2-9: Medical/Surgical History – All Subjects | 38 |
| Listing 16.2-10: Study Drug Administration – All EXPAREL Subjects | |
| Listing 16.2-11.1: All Adverse Events – All Subjects | 40 |
| Listing 16.2-11.2.1: All Treatment Emergent Adverse Events – All Subjects | 41 |
| Listing 16.2-11.2.2: All Treatment Emergent Adverse Events Related to Study Drug – All Subjects | 42 |
| Listing 16.2-11.3.1: All Serious Adverse Events – All Subjects | 43 |
| Listing 16.2-11.3.2: All Non-serious Adverse Events – All Subjects | 44 |
| Listing 16.2-11.4.1: All Treament Emergent Serious Adverse Events – All Subjects | 45 |
| Listing 16.2-11.4.2: All Treatment Emergent Non-serious Adverse Events – All Subjects | 46 |
| Listing 16.2-11.5: All Treament Emergent Study Drug Related Serious Adverse Events – All Subjects | 47 |
| Listing 16.2-12: Vital Signs – All Subjects | 48 |
| Listing 16.2-13: Numeric Rating Scale (NRS) Pain Intensity Score – All Subjects | 49 |
| Listing 16.2-14: Opioid Related Symptoms Distress Scale (ORSDS) - All Subjects | 50 |
| Listing 16.2-15: BPI-sf – All Subjects | 51 |
| Listing 16.2-16: Health Outcomes Assessments – MPADSS - All Subjects | 52 |
| Listing 16.2-17: Health Outcomes Assessments- Discharge Disposition – All Subjects | 53 |
| Listing 16.2-18.1: Phone Call / In Person Visit Day 14 (Pain Visits) - All Subjects | 54 |
| Listing 16.2-18.2: Phone Call / In Person Visit Day 14 (Medication)- All Subjects | 55 |
| Listing 16.2-19.1: Phone Call / In Person Visit Day 30 (Pain Visits) - All Subjects | 56 |
| Listing 16.2-19.2: Phone Call / In Person Visit Day 30 (Medications) - All Subjects | 57 |
| Listing 16.2-20.1: Multimodal Pain Medication – Pre-Operative – All Subjects | 58 |

| 59 |
|----|
| 60 |
| 61 |
| 62 |
| 63 |
| 64 |
| 65 |
| 66 |
| 67 |

| 402-C-413 | Statistical Analysis Plan |
|-----------------------------|---------------------------|
| acira Pharmaceuticals, Inc. | $EXPAREL^{\circledR}$ |

(Page X of Y) Pacira Pharmaceuticals, Inc. EXPAREL

402-C-413

Cohort: cohort; TREATMENT: treatment-name

Listing 16.2-1.1: Subject Disposition- All Subjects

| Additional Early<br>Termination<br>Details | XXXXXXX |
|----------------------------------------------|-------------|
| If Other,<br>Specify | XXXXX |
| Primary Reason<br>for Early<br>Termination | XXXXXX |
| End of<br>Study<br>Status | XXXXXXXX |
| Date of<br>Last Contact | DDMONYYY |
| Date of<br>the Start<br>of the<br>Last Visit | DDMONYYYY |
| Site Subject | XXX XX-YYYY |
| S<br>t<br>t | XXX |

Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH: MM

Program: program\_name

19 October 2020 21 of 68CONFIDENTIAL

| Pacira Pharmaceuticals, EXPAREL Site Subject Da | | | | Statistical Analysis Plan |
|---|---|---|---|---|
| Subject | Inc. | (Page X of Y) | | 402-C-413 |
| Subject | Listing 16.2-<br>Cohort: cohor | Listing 16.2-2: Enrollment- All Subjects Cohort: cohort; TREATMENT: treatment-name | .l Subjects<br>atment-name | |
| | Informed Consent Is t<br>Date (Day) E | Is the Subject<br>Enrolled? | <pre>Enrollment Date/Time (Day)</pre> | Enrollment Cohort |
| XXX XX-YYYY DDMC | DDMONYYYY (XX) | XXX | DDMONYYYYTHH:MM (XX) | XXXXX |

Program: program\_name Source: list SAS datasets used to create table SAS X.Y

DDMONYYYYTHH: MM

402-C-413 Statistical Analysis Plan Pacira Pharmaceuticals, Inc.  $EXPAREL^{\circledast}$ 

402-C-413 (Page X of Y) Pacira Pharmaceuticals, Inc. EXPAREL

Listing 16.2-3: Inclusion/ Exclusion Criteria- Failures Subjects

Cohort: -; Treatment: SCREEN FAILURES

| Criteria ID Failed | XXXXXXXX, XXXXXXXXX |
|------------------------------------|---------------------|
| Protocol Version<br>Enrolled Under | Version 1 |
| Informed Consent Date | DDMONYYYY |
| Site Subject | XX-XX-XX |
| Site | XXX |

DDMONYYYYTHH: MM Program: program\_name Source: list SAS datasets used to create table SAS X.Y

for example. Programmer Note: column "Criteria ID Failed" should read "Inclusion 09"

progra

Pacira Pharmaceuticals, Inc.  $\text{EXPAREL}^{\circledR}$ 

Statistical Analysis Plan

Pacira Pharmaceuticals, Inc. EXPAREL

402-C-413

Listing 16.2-4.1: Demographics - All Subjects Cohort: cohort; TREATMENT: treatment-name;

(Page X of Y)

| | XXXX | XXXX |
|-----------|-----------|-----------|
| Race | XXXXX | XXXXX |
| Ethnicity | XXXXXXXXX | XXXXXXXXX |
| Sex | × | × |
| Age (yrs) | XX | XX |
| DOB | DDMONYYYY | DDMONYYYY |
| Initials | AMZ | AMZ |
| Subject | XX-XXX | XX-YYYY |
| Site | XXX | XXX |

DDMONYYYYTHH: MM Program: program\_name Source: list SAS datasets used to create table SAS X.Y

Note to programmer: List all races checked. If race is 'other' then race should be 'Other: other-specifytext'. Statistical Analysis Plan

402-C-413

(Page X of Y) Pacira Pharmaceuticals, Inc.

EXPAREL

Listing 16.2-4.2: Demographics - Screen Failures
Cohort: cohort; TREATMENT: Screen Failures;

| Site | Subject | Initials | DOB | Age<br>(yrs) | Sex | Ethnicity | Race |
|---|---|---|---|---|---|---|---|
| | XX-YYYX | AMZ | DDMONYYYY | XX | × | XXXXXXXX | XXXXXXXXX |
| | XX-YYYY | AMZ | DDMONYYYY | XX | × | XXXXXXXXX | XXXXXXXXX |

Source: list SAS datasets used to create table

DDMONYYYYTHH: MM

Program: program\_name

SAS X.Y

Note to programmer: List all races checked. If race is 'other' then race should be 'Other: other-specifytext'.

Pacira Pharmaceuticals, Inc.

EXPAREL

402-C-413

(Page X of Y)

Listing 16.2-4.3: Demographics - Subject Enrolled but No Surgery Cohort: cohort; TREATMENT: Screen Failures;

| XXXXXXXXX | XXXXXXXXX |
|-----------|--------------------------|
| XXXXXXXXX | XXXXXXXXX |
| × | × |
| XX | XX |
| DDMONYYYY | DDMONYYYY |
| AMZ | AMZ |
| XX-XXXX | XX-YYYY |
| XXX | XXX |
| | XX-YYYY X XXXXXXXXX X XX |

Source: list SAS datasets used to create table

SAS X.Y

Program: program\_name

DDMONYYYYTHH: MM

Note to programmer: List all races checked. If race is 'other' then race should be 'Other: other-specifytext'.

Pacira Pharmaceuticals, Inc. EXPAREL

402-C-413 (Page X of Y)

Listing 16.2-5.1: Baseline Characteristics (Survey of Pain Attitudes (SOPA))- All Subjects Cohort: cohort; TREATMENT: treatment-name

| Site | Subject | Date (Day) | Data Type | Data |
|---|---|---|---|---|
| XXX | XX-XXXX | DDMONYYYY (XX) | Q1: There is little I can do to ease my pain | 0 = This is very untrue for me |
| | | | Q2: My pain does not stop me from leading a physically active life | <pre>0 = This is very untrue for<br/>me</pre> |
| | | | Q3: The pain I feel is a sign that damage is being done | <pre>0 = This is very untrue for<br/>me</pre> |
| | | | Q4: There is a connection between my emotions and my pain level | <pre>0 = This is very untrue for<br/>me</pre> |
| | | | Q5: I will probably always have to take pain medications | <pre>0 = This is very untrue for<br/>me</pre> |
| | | | Q6: When I am hurting, I deserve to be treated with care and concern | <pre>0 = This is very untrue for<br/>me</pre> |
| | | | Q7: I trust that doctors can cure my pain | <pre>0 = This is very untrue for<br/>me</pre> |

Source: list SAS datasets used to create listing

SAS X.Y

Program: program\_name

DDMONYYYYTHH: MM

Programmer Note: For column "Data Type" please display as verbatim in the shell not as what is presented in QS. QSTEST

Pacira Pharmaceuticals, Inc. EXPAREL

(Page X of Y)

402-C-413

Listing 16.2-5.2: Baseline Characteristics (Hospital Anxiety and Depression Score (HADS))- All Subjects Cohort: cohort; TREATMENT: treatment-name

| Site | Subject | Date (Day) | Data Type | Data |
|---|---|---|---|---|
| XXX | XXX-XXX | DDMONYYYY (XX) | (A) I feel tense or 'wound up' | Very often |
| | | | (D) I still enjoy the things I used to enjoy | Very often |
| | | | | Very often |
| | | | thing awful is about to happen | |
| | | | <ul><li>(D) I can laugh and see the funny side of<br/>things</li></ul> | Very often |
| | | | (A) Worrying thoughts go through my mind | Very often |
| | | | (D) I feel cheerful | Very often |
| | | | (A) I can sit at ease and feel relaxed | Very often |
| | | | (D) I feel as if I am slowed down | Very often |
| | | | (A) I get a sort of frightened feeling like "butterflies" in the stomach | Very often |
| | | | (D) I have lost interest in my appearance | Very often |
| | | | (A) I feel restless as if I have to be on the move | Very often |
| | | | (D) I look forward with enjoyment of things | Very often |
| | | | (A) I get sudden feelings of panic | Very often |
| | | | (D) I can enjoy a good book or radio or TV<br>Program | Very often |
| | | | Total Score Anxiety | 0 |
| | | | Total Score Depression | 6 |

Source: list SAS datasets used to create listing

SAS X.Y

DDMONYYYYTHH:MM

Program:program\_name

Programmer Note: For column "Data Type" please display as verbatim in the shell not as what is presented in OS. OSTEST

| Pacira Pharmaceuticals, Inc. | 402-C-41 |
|------------------------------|--------------------------|
| EXPAREL® | Statistical Analysis Pla |

402-C-413 (Page X of Y) Pacira Pharmaceuticals, Inc. EXPAREL

Listing 16.2-5.3: Baseline Characteristics (5-Item Opioid Compliance Checklist (OCC) - All Subjects Cohort: cohort; TREATMENT: treatment-name

| Site | Site Subject | Date (Day) | Data Type | Data |
|---|---|---|---|---|
| XXX | XX-XXX | DDMONYYYY (XX) | XX) Over the past month have you: | |
| | | | 1. Lost or misplaced your opioid medications? | Yes |
| | | | 2. Run out of your pain medication early? | Yes |
| | | | 3. Missed any scheduled medical appointments? | Yes |
| | | | 4. Used any illegal or unauthorized substances? | Yes |
| | | | 5. Been completely honest about your personal drug | Yes |
| | | | use? | |

Source: list SAS datasets used to create table

SAS X.Y

Program:program\_name

DDMONYYYYTHH: MM

Programmer Note: For column "Data Type" please display as verbatim in the shell not as what is presented in QS.QSTEST

402-C-413 Statistical Analysis Plan

402-C-413

(Page X of Y) Pacira Pharmaceuticals, Inc EXPAREL

Pacira Pharmaceuticals, Inc.  $EXPAREL^{\circledast}$ 

Listing 16.2-6.1: Pregnancy test- All Female Subects
Cohort: cohort; TREATMENT: treatment-name

| Test Result | XXXXX |
|-------------------------------------------|--------|
| If Yes, Was Urine<br>Pregnancy Test done? | × |
| Is subject of child bearing potential? | × |
| Subject | XX-XXX |
| Site | XXX |

DDMONYYYYTHH: MM Program: program\_name Source: list SAS datasets used to create table SAS X.Y

Pacira Pharmaceuticals, Inc EXPAREL

(Page X of Y)

402-C-413

Listing 16.2-6.2: Pregnancy test- Female Screen Fails

| E () | 4 |
|------------------------------------------|----------------------|
| If Yes, Was Urine | Pregnancy Test done? |
| Is subject of child bearing | potential? |
| Subject | |
| ()<br>+<br>-r | טדרת |

XX-YYYY  $\times \times \times$ 

 $\bowtie$ 

 $\bowtie$ 

XXXXX

Source: list SAS datasets used to create table

SAS X.Y

Program: program\_name

DDMONYYYYTHH: MM

402-C-413

Pacira Pharmaceuticals, Inc.  $\mathsf{EXPAREL}^{\scriptscriptstyle{\circledR}}$ 

Statistical Analysis Plan

Pacira Pharmaceuticals, Inc. EXPAREL

(Page X of Y)

402-C-413

Listing 16.2-7.1: Admission and Discharge- Post-Anesthesia Care Unit (PACU) - All Subjects Cohort: cohort; TREATMENT: treatment-name

| | Subject | Admission<br>Date/Time (Day) | Discharge<br>Date/Time (Day) | Total length of stay (hours) |
|---|---|---|---|---|
| X | XX-XXX | DDMONYYYYTHH:MM (XX) | DDMONYYYYTHH:MM (XX) | X.XXX |

Source: list SAS datasets used to create table

SAS X.Y

Program: program\_name

DDMONYYYYTHH: MM

Programmer Note: For column "Total length of stay (hours)" please populate with the numeric number not as PODIIH24M as displayed in SDIM.HO.HODUR

402-C-413

Pacira Pharmaceuticals, Inc.  $EXPAREL^{\circledR}$ 

Statistical Analysis Plan

(Page X of Y)

Protocol: 402-C-413

Pacira Pharmaceuticals EXPAREL

Listing 16.2-7.2: Admission and Discharge - Surgical Facility - All Subjects

Cohort: cohort; TREATMENT: treatment-name

hospital/facility Total length of stay in (hours) stay in step-down Total length of (hours) Date/ Time (Day) Discharge Date/ Time (Day) Admission Subject Site

 $\times$ 

 $\times$ 

DDMONYYYYTHH:MM (XX)

DDMONYYYYTHH: MM (XX)

XX-YYYY

XXX

DDMONYYYYTHH: MM Source: list SAS datasets used to create table

SAS X.Y

Program: program\_name

Programmer Note: For column "Total length of stay in hospital/facility (hours)" please populate with the numeric number not as PODT1H24M as displayed in SDTM.HO.HODUR Pacira Pharmaceuticals, Inc. EXPAREL  $^{\circledR}$ 

402-C-413 (Page X of Y) Pacira Pharmaceuticals, Inc. EXPAREL

Listing 16.2-8.1: Surgery Characteristics- Procedure - All Subjects Cohort: cohort; TREATMENT: treatment-name

| • | |
|---|---|
| Incision<br>Length (cm) | m |
| Surgery<br>Performed by | XXX |
| Procedure Name | XXXXXX/ Subtypes |
| <pre>Start Date/ Time (Day)/ End Date/Time (Day)/ Duration [1]</pre> | DDMONYYYYTHH:MM (XX)/ DDMONYYYYTHH:MM (XX)/ XXXX |
| Subject | XX-XXX |
| Site | XXX |

[1] Duration of surgery is calculated as the difference between the end of surgery and start of surgery times and reported in hours

Source: list SAS datasets used to create table

SAS X.Y

Program: program\_name

DDMONYYYYTHH: MM

Statistical Analysis Plan Pacira Pharmaceuticals, Inc. EXPAREL  $^{\otimes}$ 

Pacira Pharmaceuticals, Inc EXPAREL

402-C-413

Listing 16.2-8.2: Surgery Characteristics- Anesthesia- All Subjects Cohort: cohort; TREATMENT: treatment-name

(Page X of Y)

| | ĸ | |
|---------------|------------|---------------|
| Type of | Anesthesia | XXXXX |
| Anesthsia | End Time | нн: им |
| Anesthsia | Start Time | нн: мм |
| Surgery Start | Date (Day) | DDMONYYY (XX) |
| Subject | | XX-XXXX |
| Site | | XXX |

Source: list SAS datasets used to create table

SAS X.Y

Program: program\_name

DDMONYYYYTHH: MM

Note to programmer: If anesthesia type is 'other' then text should read 'other: specify-text'.

402-C-413

Pacira Pharmaceuticals, Inc.  $EXPAREL^{\circledast}$ 

Pacira Pharmaceuticals, Inc. EXPAREL

(Page X of Y)

| If Yes, Harvest Site | Other: XXXXXX |
|--------------------------|----------------|
| Was an Autograft Taken? | Yes |
| Surgery Start Date (Day) | DDMONYYYY (XX) |
| Subject | XX-XXXX |
| Site | XXX |

Source: list SAS datasets used to create table

SAS X.Y

Program: program\_name

DDMONYYYYTHH: MM
Pacira Pharmaceuticals, Inc.  $\text{EXPAREL}^{\circledR}$ 

Statistical Analysis Plan

Pacira Pharmaceuticals, Inc. EXPAREL

402-C-413

Listing 16.2-8.4: Surgery Characteristics-Prior Staged Procedure - All Subjects Cohort: cohort; TREATMENT: treatment-name

(Page X of Y)

| Stop Date/Time (Day) |
|-------------------------------------------|
| Start Date/Time (Day) |
| Staged Procedure Type |
| Surgery part<br>of a staged<br>procedure? |
| Site Subject |

DDMONYYYYTHH:MM (XX) DDMONYYYYTHH:MM (XX) XXXXXXXX  $\times \times \times$ XX-YYYY XXX

Source: list SAS datasets used to create table

SAS X.Y

Program: program\_name

DDMONYYYYTHH: MM

402-C-413 Statistical Analysis Plan Pacira Pharmaceuticals, Inc. EXPAREL®

(Page X of Y) Pacira Pharmaceuticals, Inc. EXPAREL

402-C-413

Listing 16.2-9: Medical/Surgical History - All Subjects

Cohort: cohort; Treatment: treatment-name

| Data | DDMONYYYY | DDMONYYYY | XXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
|---|---|---|---|---|---|
| Data Type | Start Date | Stop Date | System Organ Class | Preferred | Verbatim |
| Medical History<br>Number | XX | | | | |
| Site Subject | XX-YYYY | | | | |
| Site | XXX | | | | |

Note: Only subjects with relevant medicial history or surgery are included in this listing.

DDMONYYYYTHH: MM Source: list SAS datasets used to create listing

SAS X.Y

Program:program\_name

pages. Insert a page break between subjects. The column "Medicial History Number" should correspond to MHSEQ Note to programmer: If condition is ongoing, put ONGOING in stop row. Do not split a condition across

| Pacira Pharmaceuticals, Inc. EXPAREL® | Statisti | 402-C-413<br>Statistical Analysis Plan |
|---|---|---|
| Pacira Pharmaceuticals, Inc.<br>EXPAREL | (Page X of Y) | 402-C-413 |
| Tisting 16 2-10. | Tisting 16 2-10. Study Drug Administration - All EXPARET. Subjects | |

LISTING 16.2-10: Study Drug Administration - All EXPAREL Subjects Cohort: cohort; TREATMENT: EXPAREL

| Study Drug<br>Administered by | XXX |
|---|---|
| Total<br>Volume (mL) | XXX |
| Start Date/Time (Day)/<br>End Date/Time (Day | DDMONYYYYTHH:MM (XX)/<br>DDMONYYYYTHH:MM (XX) |
| Case Obs<br>Correctly? | XXX |
| Subject | XX-XXX |
| Site | XXX |

Note: Only subjects in Cohort 3 were administered EXPAREL.

Source: list SAS datasets used to create table

DDMONYYYYTHH: MM

Program: program\_name

SAS X.Y

Note to programmer: If Not Done is checked then text should read 'Not Done: reason-text'.

| Pacira Pharmaceuticals, Inc. (Page X of |
|-----------------------------------------|

Listing 16.2-11.1: All Adverse Events - All Subjects

EXPAREL

Cohort: cohort; Treatment: treatment-name

| <br>+<br>+ | ب<br>1<br>1<br>1<br>1<br>1<br>1 | TEN | פרייד ב + בר | |
|---|---|---|---|---|
| ט<br>ר | Sab Jace | 1 | | שמרמ |
| XXX | XX-YYYY | Z | Start Date/ Time (Day) | DDMONYYYYTHH:MM (XX) |
| | | | Stop Date/ Time (Day) | DDMONYYYYTHH:MM (XX) |
| | | | AE Number | × |
| | | | System Organ Class | XXXXXXXXXXXXXXX |
| | | | Preferred | XXXXXXXXXXXXXXXXXX |
| | | | Verbatim | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | | Severity | XXXXXXXX |
| | | | Relationship to Study<br>Drug | XXXXXXX |
| | | | Action Taken with Subject | XXXXXXXXXXXXXXXXXX |
| | | | Outcome | XXXXXXXXXXXXX |
| | | | Serious | XXX |
| | | | Serious Cause(s) | XXXXXXXXXXX |
| | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

TEAE: Treatment-emergent AE (Y=TEAE/N=Not TEAE)

Source: list SAS datasets used to create listing

DDMONYYYYTHH: MM

Program: program\_name

SAS X.Y

402-C-413 Statistical Analysis Plan Pacira Pharmaceuticals, Inc. EXPAREL®

Protocol: 402-C-413 (Page X of Y) Pacira Pharmaceuticals EXPAREL

Listing 16.2-11.2.1: All Treatment Emergent Adverse Events - All Subjects

Cohort: cohort; Treatment: treatment-name

| Site | Subject | Data Type | Data |
|---|---|---|---|
| XXX | XX-YYYY | Start Date/ Time (Day) | DDMONYYYYTHH:MM (XX) |
| | | Stop Date/ Time (Day) | DDMONYYYYTHH:MM (XX) |
| | | AE Number | × |
| | | System Organ Class | XXXXXXXXXXXXXXXX |
| | | Preferred | XXXXXXXXXXXXXXXXXX |
| | | Verbatim | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | Severity | XXXXXXXX |
| | | Relationship to Study<br>Drug | XXXXXXX |
| | | Action Taken with Subject | XXXXXXXXXXXXXXXXXX |
| | | Outcome | XXXXXXXXXXXX |
| | | Serious | XXX |
| | | Serious Cause(s) | XXXXXXXXXXXX |
| | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

TEAE: Treatment-emergent AE (Y=TEAE/N=Not TEAE)

Source: list SAS datasets used to create listing

DDMONYYYYTHH: MM

program\_name

SAS X.Y

Statistical Analysis Plan 402-C-413 Pacira Pharmaceuticals, Inc. EXPAREL® Protocol: 402-C-413  $\vec{\lambda}$ (Page X of Pacira Pharmaceuticals, Inc. EXPAREL

Listing 16.2-11.2.2: All Treatment Emergent Adverse Events Related to Study Drug - All Subjects

Cohort: cohort; Treatment: treatment-name

XXXXXXXXXXXXXXXXXXX XXXXXXXXXXXXXXXXX XXXXXXXXXXXXXXXXXX DDMONYYYYTHH: MM (XX) (XX) MM: HHIXXXXNOWQQ XXXXXXXXXXXXXXXX XXXXXXXXXXXX XXXXXXXXXXXXX XXXXXXXX XXXXXXXX Data  $\times \times \times$ Action Taken with Subject Start Date/ Time (Day) Relationship to Study Stop Date/ Time (Day) System Organ Class Serious Cause(s) Verbatim Preferred Data Type AE Number Severity Outcome Serious Drug Subject XXX-XX Site XXX

TEAE: Treatment-emergent AE (Y=TEAE/N=Not TEAE)

Source: list SAS datasets used to create listing

DDMONYYYYTHH: MM

program\_name

SAS X.Y

| 402-C-413 | Statistical Analysis Plan |
|-------------------------|---------------------------|
| , Inc. | |
| Pacira Pharmaceuticals, | EXPAREL® |

Listing 16.2-11.3.1: All Serious Adverse Events - All Subjects Cohort: cohort; Treatment: treatment-name

| Site | Subject | TEAE | TEAE Data Type | Data |
|---|---|---|---|---|
| XXX | XX-YYYY | Z | Start Date/ Time (XX) | DDMONYYYYTHH:MM (XX) |
| | | | Stop Date/ Time (XX) | DDMONYYYYTHH:MM (XX) |
| | | | AE Number | $\times$ |
| | | | System Organ Class | XXXXXXXXXXXXXXX |
| | | | Preferred | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | | Verbatim | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | | Severity | XXXXXXXX |
| | | | Relationship to Study<br>Drug | XXXXXXXX |
| | | | Action Taken | XXXXXXXXXXXXXXXXXX |
| | | | Outcome | XXXXXXXXXXXXX |
| | | | Serious | XXX |
| | | | Serious Cause(s) | XXXXXXXXXXXXX |
| | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

TEAE: Treatment-emergent AE (Y=TEAE/N=Not TEAE)

Source: list SAS datasets used to create listing

DDMONYYYYTHH:MM program\_name

SAS X.Y

| 402-C-413 | itistical Analysis Plan |
|-----------------------------|-------------------------|
| | Sta |
| acira Pharmaceuticals, Inc. | EXPAREL® |

Listing 16.2-11.3.2: All Non-serious Adverse Events - All Subjects

Cohort: cohort; Treatment: treatment-name

| Site | Subject | TEAE | Data Type | Data |
|---|---|---|---|---|
| XXX | XX-YYYY | Z | Start Date/ Time (XX) | DDMONYYYYTHH:MM (XX) |
| | | | Stop Date/ Time (XX) | DDMONYYYYTHH:MM (XX) |
| | | | AE Number | × |
| | | | System Organ Class | XXXXXXXXXXXXXXXX |
| | | | Preferred | XXXXXXXXXXXXXXXXXX |
| | | | Verbatim | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | | Severity | XXXXXXXX |
| | | | Relationship to Study<br>Drug | XXXXXXXX |
| | | | Action Taken | XXXXXXXXXXXXXXXXXX |
| | | | Outcome | XXXXXXXXXXXXX |
| | | | Serious | XXX |
| | | | Serious Cause(s) | XXXXXXXXXXX |
| | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

TEAE: Treatment-emergent AE (Y=TEAE/N=Not TEAE)

Source: list SAS datasets used to create listing

DDMONYYYYTHH:MM program\_name

SAS X.Y

402-C-413 Statistical Analysis Plan Pacira Pharmaceuticals, Inc.  $EXPAREL^{\circledR}$ 

Protocol: 402-C-413 (Page X of Y) Pacira Pharmaceuticals EXPAREL, Inc.

Listing 16.2-11.4.1: All Treament Emergent Serious Adverse Events - All Subjects Cohort: cohort; Treatment: treatment-name

| Site | Subject | Data Type | Data |
|---|---|---|---|
| XXX | XX-YYYY | Start Date/ Time (XX) | DDMONYYYYTHH:MM (XX) |
| | | Stop Date/ Time (XX) | DDMONYYYYTHH:MM (XX) |
| | | AE Number | × |
| | | System Organ Class | XXXXXXXXXXXXXXXX |
| | | Preferred | XXXXXXXXXXXXXXXXX |
| | | Verbatim | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | Severity | XXXXXXXX |
| | | Relationship to Study<br>Drug | XXXXXXXX |
| | | Action Taken | XXXXXXXXXXXXXXXXXX |
| | | Outcome | XXXXXXXXXXXXX |
| | | Serious | XXX |
| | | Serious Cause(s) | XXXXXXXXXXXX |
| | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

TEAE: Treatment-emergent AE (Y=TEAE/N=Not TEAE)

Source: list SAS datasets used to create listing

DDMONYYYYTHH: MM

program\_name

SAS X.Y

402-C-413 Statistical Analysis Plan Pacira Pharmaceuticals, Inc.  $EXPAREL^{\circledR}$  Protocol: 402-C-413 (Page X of Y) Pacira Pharmaceuticals, Inc. EXPAREL

Listing 16.2-11.4.2: All Treatment Emergent Non-serious Adverse Events - All Subjects Cohort: cohort; Treatment: treatment-name

| Site | Subject | Data Type | Data |
|---|---|---|---|
| XXX | XX-YYYY | Start Date/ Time (XX) | DDMONYYYYTHH:MM (XX) |
| | | Stop Date/ Time (XX) | DDMONYYYYTHH:MM (XX) |
| | | AE Number | × |
| | | System Organ Class | XXXXXXXXXXXXXXXX |
| | | Preferred | XXXXXXXXXXXXXXXXXX |
| | | Verbatim | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | Severity | XXXXXXX |
| | | Relationship to Study<br>Drug | XXXXXXX |
| | | Action Taken | XXXXXXXXXXXXXXXXXX |
| | | Outcome | XXXXXXXXXXXX |
| | | Serious | XXX |
| | | Serious Cause(s) | XXXXXXXXXXXX |
| | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

TEAE: Treatment-emergent AE (Y=TEAE/N=Not TEAE)

Source: list SAS datasets used to create listing

DDMONYYYYTHH: MM

program\_name

SAS X.Y

Listing 16.2-11.5: All Treament Emergent Study Drug Related Serious Adverse Events - All Subjects Cohort: cohort; Treatment: treatment-name

| Site | Subject | Data Type | Data |
|---|---|---|---|
| XXX | XX-YYYY | Start Date/ Time (XX) | DDMONYYYYTHH:MM (XX) |
| | | Stop Date/ Time (XX) | DDMONYYYYTHH:MM (XX) |
| | | AE Number | × |
| | | System Organ Class | XXXXXXXXXXXXXXXX |
| | | Preferred | XXXXXXXXXXXXXXXXXX |
| | | Verbatim | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | Severity | XXXXXXX |
| | | Relationship to Study<br>Drug | XXXXXXX |
| | | Action Taken | XXXXXXXXXXXXXXXXXX |
| | | Outcome | XXXXXXXXXXXX |
| | | Serious | XXX |
| | | Serious Cause(s) | XXXXXXXXXXXX |
| | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

TEAE: Treatment-emergent AE (Y=TEAE/N=Not TEAE)

Source: list SAS datasets used to create listing

DDMONYYYYTHH:MM program\_name

SAS X.Y

Listing 16.2-12: Vital Signs - All Subjects Cohort: cohort; TREATMENT: treatment-name

| Date/Time (Day) Height Weight BMI (kg) | DDMONYYYYTHH:MM (XX) XX XX XX XX | XX | | 7777 |
|---|---|---|---|---|
| Date/Time (Day) | DDMONYYYYTHH:MM (XX) | | DDMONYYYYTHH:MM (XX) | |
| Done? | Yes | Yes | Yes | |
| Subject | XX-XXXX | XX - XXXX | XX-YYYY | |
| Site | XXX | XXX | XXX | |

DDMONYYYYTHH: MM Program:program\_name Source: list SAS datasets used to create table SAS X.Y

Note to programmer: If Not Done is checked then text should read 'Not Done: reason-text'. If data is missing populate with "-".

Listing 16.2-13: Numeric Rating Scale (NRS) Pain Intensity Score - All Subjects

Cohort: cohort; TREATMENT: treatment-name

| Site | Subject | Time Point / Asleep<br>During Time Point [1] | Date/Time (Day) | NRS Pain<br>Intensity Score |
|---|---|---|---|---|
| XXX | XX-XXX | Screening | DDMONYYYYTHH:MM (XX) | I |
| | | 48 hours / No | DDMONYYYYTHH:MM (XX) | XXX |
| | | Discharge | DDMONYYYYTHH:MM (XX) | XXX |
| | | 14 days | DDMONYYYYTHH:MM (XX) | XXX |

 $\overline{72}$  hours. I [1] Asleep During Time Point only used for schelduled 6

Source: list SAS datasets used to create table

SAS X.Y

DDMONYYYYTHH: MM

Program: program\_name

subject is considered to be asleep during an assessment if SDTM.QS.qscat="NRS-R Pain Intensity" Note to programmer: Include all NRS scores. For colum "Time Point / Asleep During Time Point [1]" a and QSREASND="ASLEEP" 402-C-413

(Page X of Y) Pacira Pharmaceuticals, Inc. EXPAREL

Listing 16.2-14: Opioid Related Symptoms Distress Scale (ORSDS) - All Subjects Cohort: cohort; TREATMENT: treatment-name

| Distress | Did # or | Have Episodes Often Severe Bother | , l | Drowsiness - Occasionally Slight A little | Concentrate N | Z | Z | Constipation N | N | Z | Z | Retching/vomiting $_{ m N}$ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Date/Time (Day) | | DDMONYYYYTHH: MM: (XX) | | | | | | | | | |
| (<br>}<br>-! | Point | )<br> | 24 hrs | | | | | | | | | |
| | Site Subject | | XXX XX-YYYY 24 hrs | | | | | | | | | |
| | Site | | XXX | | | | | | | | | |

Note to programmer: Add in all applicable visits.

SAS X.Y

Program: program\_name

Pacira Pharmaceuticals, Inc.  $EXPAREL^{\circledast}$ 

Pacira Pharmaceuticals EXPAREL

(Page X of Y)

402-C-413

Listing 16.2-15: BPI-sf - All Subjects Cohort: cohort; TREATMENT: treatment-name

| Data | Yes | Front leg, | Back Ley<br>Front Leg | 1 | | 5 | ĸ | | 7 | | | | 2 | | <sub>8</sub> | | 4 | | 2 | | <b>⊢</b> | | $\vdash$ | | 8 | | DDMONYYYYTHH: MM |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Data Type | Have you had pain, other than everyday pain kinds of pain today? | | Area where it hurts the most | e your pain that descr | vorst in the last 24 hours | Rate your pain that describes your pain at<br>its least in the last 24 hours | pain that descr | average | Rate your pain that describes your pain | right now | In the last 24 hours, how much relief have | pain medications provided? (Percentage) | 24 hours | ered with: General | During the past 24 hours pain has | interfered with: Mood | | interfered with: Walking Abililty | During the past 24 hours pain has | interfered with: Normal Work | During the past 24 hours pain has | interfered with: Relationships | During the past 24 hours pain has | interfered with: Sleep | During the past 24 hours pain has | ered with: Enjoymer | table |
| Date of<br>Assessment | DDMONYYYYTHH: MM | | | | | | | | | | | | | | | | | | | | | | | | | | used to create ta |
| Timepoint | Screening | | | | | | | | | | | | | | | | | | | | | | | | | | datasets |
| Subject | XXX-XX | | | | | | | | | | | | | | | | | | | | | | | | | | : list SAS |
| Site | XXX | | | | | | | | | | | | | | | | | | | | | | | | | | Source: |

SAS X.Y

402-C-413

(Page X of Y) Pacira Pharmaceuticals, Inc. EXPAREL

Listing 16.2-16: Health Outcomes Assessments - MPADSS - All Subjects Cohort: cohort; TREATMENT: treatment-name

| Site | Subject | Subject Timepoint Done? | Done? | Date/ Time (Day) | Data Type | Data |
|---|---|---|---|---|---|---|
| XXX | XX-XXX | XX-YYYY 24 Hours | Yes | DDMONYYYYTHH:MM (XX) | Vital Signs | 2 = <=20% of preoperative value |
| | | | | | Ambulation | <pre>2 = Steady gait/no dizziness</pre> |
| | | | | | Nausea/Vomiting | 2 = Minimal |
| | | | | | Pain | 2 = Minimal |
| | | | | | Surgical Bleeding | 2 = Minimal |
| | | | | | Score | 10 |
| ××× | XX-YYYY | XX-YYYY 48 Hours | No, XX | DDMONYYYYTHH:MM (XX) | | |

MPADSS= Modified Post-Anesthesia Discharge Scoring System;

Source: list SAS datasets used to create table

DDMONYYYYTHH: MM

SAS X.Y

Note to programmer: If Not Done is checked then text should read 'Not Done: reason-text'.

Pacira Pharmaceuticals, Inc.

**EXPAREL®** 

Statistical Analysis Plan

Pacira Pharmaceuticals, Inc. EXPAREL

402-C-413

Listing 16.2-17: Health Outcomes Assessments- Discharge Disposition - All Subjects Cohort: cohort; TREATMENT: treatment-name

(Page X of Y)

| Site | Subject | Where will the Subject be Discharged? |
|------|---------|---------------------------------------|
| XXX | XX-YYYY | Home |
| XXX | XX-YYYY | Home |
| XXX | XXX-XX | Home |
| × | XX-XXXX | Home |

Source: list SAS datasets used to create table

SAS X.Y

Program: program\_name

DDMONYYYYTHH: MM

Programmer Note: if column "Where will the Subject be Discharged?" is Other, it should read "Other:text".

Pacira Pharmaceuticals, Inc. **EXPAREL®** 

Statistical Analysis Plan

402-C-413

(Page X of Y) Pacira Pharmaceuticals, Inc EXPAREL

Listing 16.2-18.1: Phone Call / In Person Visit Day 14 (Pain Visits) - All Subjects Cohort: cohort; TREATMENT: treatment-name

| | | | | | , |
|---|---|---|---|---|---|
| If Yes,<br>Number<br>of<br>Pain-<br>related<br>Visits | XXX | XXX | XXX | XXX | XXX |
| Any Unscheduled<br>Pain-Related<br>Visits Since<br>Discharge? | XXX | XXX | XXX | XXX | XXX |
| How Many Times<br>Called<br>Physician About<br>Pain Related to<br>Your Surgery? | XXX | XXX | XXX | XXX | XXX |
| Date of Visit<br>(Day) | DDMONYYY (XX) | DDMONYYYY (XX) | DDMONYYYY (XX) | DDMONYYY (XX) | DDMONYYYY (XX) |
| Phone Call<br>or In Person<br>Visit? | XXX | XXX | XXX | XXX | XXX |
| Completed? | XXX | XXX | XXX | XXX | XXX |
| Subject | XX-YYYY | XX-XXX | XX-YYYY | XX-YYYY | XX-YYYY |
| Site | XXX | XXX | ×× | XXX | XXX |

Source: list SAS datasets used to create table

SAS X.Y

Program: program\_name

DDMONYYYYTHH: MM

Note to programmer: If Was Day 14 Visit Completed? is 'No' then text should read 'No: reason-text'.

Pacira Pharmaceuticals, Inc. EXPAREL®

Statistical Analysis Plan

402-C-413 (Page X of Y) Pacira Pharmaceuticals, Inc. EXPAREL

Listing 16.2-18.2: Phone Call / In Person Visit Day 14 (Medication) - All Subjects Cohort: cohort; TREATMENT: treatment-name

| mber of<br>quests | | | | | |
|---|---|---|---|---|---|
| If Yes, Number of<br>Refill Requests | XXX | XXX | XXX | XXX | XXX |
| Any Requests for<br>Refills for Opioid<br>Medication? | ××× | XXX | XXX | XXX | XXX |
| Date of Visit<br>(Day) | DDMONYYYY (XX) | DDMONYYYY (XX) | DDMONYYYY (XX) | DDMONYYYY (XX) | DDMONYYYY (XX) |
| Phone Call or In Date of Visit<br>Person Visit? (Day) | ×× | XXX | XXX | XXX | XXX |
| Completed? | XXX | XXX | XXX | XXX | ×× |
| Site Subject | XX-YYYY | XX-YYYY | XX-YYYY | XX-YYY | XX-XXXX |
| Site | XXX | XXX | XXX | XXX | XXX |

Source: list SAS datasets used to create table

DDMONYYYYTHH: MM

program\_name

SAS X.Y

Note to programmer: If Was Day 14 Visit Completed? is 'No' then text should read 'No: reason-text'.

402-C-413

(Page X of Y) Pacira Pharmaceuticals, Inc EXPAREL

Listing 16.2-19.1: Phone Call / In Person Visit Day 30 (Pain Visits) - All Subjects Cohort: cohort; TREATMENT: treatment-name

| Was Phone<br>Call Made to<br>the Subject? | Date of Phone<br>Contact (Day) | Any Hospital/ Facility Readmissions Since Discharge? (Number) | If Yes, Of the Total Readmissions, How Many Were Related to Pain | Any ED Visits<br>Since Subject<br>Discharge?<br>(Number) |
|---|---|---|---|---|
| XXX | DDMONYYYY (XX) | XXX (xx) | XXX | XXX (xx) |
| | DDMONYYYY (XX) | XXX (xx) | XXX | XXX (xx) |
| | DDMONYYYY (XX) | XXX (xx) | XXX | XXX (xx) |
| | DDMONYYYY (XX) | XXX (xx) | XXX | XXX (xx) |
| | DDMONYYYY (XX) | XXX (xx) | XXX | XXX (xx) |

DDMONYYYYTHH: MM Source: list SAS datasets used to create table SAS X.Y

Note to programmer: If Was Day 30 Visit Completed? is 'No' then text should read 'No: reason-text'.

Program: program\_name

402-C-413 (Page X of Y) Pacira Pharmaceuticals, Inc. EXPAREL

Listing 16.2-19.2: Phone Call / In Person Visit Day 30 (Medications) - All Subjects

| ) | |
|---|-------------------------------------------|
| 1 | |
| | Cohort: cohort; TREATMENT: treatment-name |
| 1 | YIMENT: |
| ) | · TREA |
| | short, |
| 1 | Cohort: cohort; |
| | Coho |
| 1 | |
| 1 | |
| 2 | |

| ing | | | | | |
|---|---|---|---|---|---|
| Currently Taking<br>Opioid<br>Medications? | XXX | XXX | XXX | XXX | XXX |
| Date of Phone Contact (Day) | (X | (× | (X | (X | (× |
| of Phon | (XX) XXXANOMOC | DMONYYYY (XX) | YYYY (XX) | YYYY (XX) | YYYY (XX) |
| | NOMQQ | DDMON | DDMONYYYY | DDMONYYYY | DDMONYYYY |
| de to the | | | | | |
| Was Phone Call Made to the<br>Subject? | XXX | XXX | XXX | XXX | XXX |
| Subject | XX-XXXX | XX-YYYY | XX-YYYY | XX-YYYY | XX-YYYY |
| Site | XXX | XXX | XXX | XXX | XXX |

Source: list SAS datasets used to create table

SAS X.Y

Program: program\_name

DDMONYYYYTHH: MM

Note to programmer: If Was Day 30 Visit Completed? is 'No' then text should read 'No: reason-text'.

402-C-413

(Page X of Y) Pacira Pharmaceuticals, Inc. EXPAREL

Listing 16.2-20.1: Multimodal Pain Medication - Pre-Operative - All Subjects Cohort: cohort; TREATMENT: treatment-name

| Φ | |
|---|---|
| Route | * * * * |
| Dose (units) | (XXXX) XX<br>(XXXX) XX<br>(XXXX) XX<br>(XXXX) XX |
| Λ) | (XX)<br>(XX)<br>(XX)<br>(XX) |
| Date/ Time (Day) | DDMONYYYYTHH:MM<br>DDMONYYYYTHH:MM<br>DDMONYYYYTHH:MM |
| Was Medication<br>Taken? | XXX<br>XXX<br>XXX |
| Medication | Tylenol (PO)<br>Gabapentin (PO)<br>Robaxin (PO)<br>Pregabalin (PO) |
| Site Subject | XX-XXXX |
| Site | XXX |

Source: list SAS datasets used to create table

SAS X.Y

Program: program\_name

DDMONYYYYTHH: MM

Note to programmer: If Mediciation is not taken then text should read 'No: reason-text'.

Pacira Pharmaceuticals, Inc. EXPAREL®

402-C-413 (Page X of Y) Pacira Pharmaceuticals, Inc. EXPAREL

Listing 16.2-20.2: Multimodal Pain Medication - Post-Operative - All Subjects Cohort: cohort; TREATMENT: treatment-name

| Site | Site Subject | Medication | Was Medication<br>Taken? | Date/ Time (Day) | Dose (units) | Route |
|---|---|---|---|---|---|---|
| XXX | XX-YYYY | Tylenol (PO) | XXX | DDMONYYYYTHH:MM (XX) | (XXXX) | XX |
| | | Gabapentin (PO) | XXX | DDMONYYYYTHH:MM (XX) | XX (XXXX) | ×× |
| | | Robaxin (PO) | XXX | DDMONYYYYTHH:MM (XX) | XX (XXXX) | XX |
| | | Pregabalin (PO) | XXX | DDMONYYYYTHH:MM (XX) | (XXXX) | XX |

DDMONYYYYTHH: MM Program: program\_name Source: list SAS datasets used to create table SAS X.Y

Note to programmer: If Mediciation is not taken then text should read 'No: reason-text'.

| Pacira Pharmaceuticals, Inc. | 402-C-413 |
|------------------------------|---------------------------|
| $EXPAREL^{\otimes}$ | Statistical Analysis Plan |

402-C-413 (Page X of Y) Pacira Pharmaceuticals, Inc. EXPAREL

Listing 16.2-20.3: Intraoperative Medications - All Subjects Cohort: cohort; Treatment: treatment-name

XXXXXXXXXXXXXXXXXXXX XXXXXXXXXXXXXXXXXXX XXXXXXXXXXXXXXXXX XXXXXXXXXXXXXXXXX XXXXXXXXXXXXXXXXXXX XXXXXXXXXXXXXXX  $\times$ DDMONYYYYTHH: MM DDMONYYYYTHH: MM XXX AE # XX, XXXXXXXX XXXXXXXX XXXXXXXX Data × 4 Medication Number Start Date/ Time Preferred Name ATC Level # End Date/ Time ATC Level Associated AE ablaVerbatim ATC Level ATC Level 1 Data Type Route Unit Dose Subject XXXX-XX Site XXX

ATC=Anatomical therapeutic class

Source: list SAS datasets used to create listing

DDMONYYYYTHH: MM

Program: program\_name

SAS X.Y

α Note to programmer: If medication has unknown end time, put 'Unknown' after date in End row. Do not split medication across pages. The AE number should correspond SDTM.AE.AESEQ 402-C-413

Statistical Analysis Plan Pacira Pharmaceuticals, Inc.  $EXPAREL^{\circledR}$ 

(Page X of Y) Pacira Pharmaceuticals, Inc. EXPAREL

Listing 16.2-20.4: Prescription Daily Pain Medications - All Subjects

Cohort: cohort; Treatment: treatment-name

Site XXX

| Subject | Data Type | Data |
|---------|-------------------|-----------------------------------------|
| XX-YYYY | Start Date/ Time | DDMONYYYYTHH:MM |
| | Medication Number | $\times$ |
| | ATC Level 1 | XXXXXXXXXXXXXXXX |
| | ATC Level 2 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | ATC Level 3 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | ATC Level 4 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | Preferred Name | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | Verbatim | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | Dose | XXXXXXXX |
| | Unit | XXXXXXXX |
| | Route | XXXXXXXX |

ATC=Anatomical therapeutic class

Source: list SAS datasets used to create listing

DDMONYYYYTHH: MM

Program: program name

SAS X.Y

Note to programmer: If medication has unknown end time, put 'Unknown' after date in End row. Do not split a medication across pages. If Unit or Route is 'Other', text should read 'Other: specify-text'. Insert a page break between subjects. 402-C-413

Statistical Analysis Plan Pacira Pharmaceuticals, Inc.  $EXPAREL^{\circledast}$ 

Pacira Pharmaceuticals, Inc. EXPAREL

(Page X of Y)

Listing 16.2-20.5: Rescue Medication - All Subjects Cohort: cohort; TREATMENT: treatment-name

| Site | Subject | Medication | Date/ Time (Day) | Dose (unit) | Route |
|---|---|---|---|---|---|
| ××× | XX-YYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMONYYYYTHH:MM (XX) DDMONYYYYTHH:MM (XX) DDMONYYYYTHH:MM (XX) | XX (mg) XX (mg) XX (mg) XX (mg) | XXXXXXX<br>XXXXXXX<br>XXXXXXX |

Source: list SAS datasets used to create table

DDMONYYYYTHH: MM

Program: program\_name

SAS X.Y

402-C-413 Statistical Analysis Plan Pacira Pharmaceuticals, Inc.  $\text{EXPAREL}^{\circledR}$ 

(Page X of Y) Pacira Pharmaceuticals, Inc. EXPAREL

402-C-413

Listing 16.2-20.6: Prior Medications - All Subjects Cohort: cohort; Treatment: treatment-name

| Data | DDMONYYYYTHH:MM | DDMONYYYYTHH:MM | × | XXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXX (XXXXXXXXX) | XXXXXXXX | XXXXXXX | XXXXXXXXXXXXXX AE # XX (or MH # XX) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Data Type | Start Date and Time | End Date and Time | Medication Number | ATC Level 1 | ATC Level 2 | ATC Level 3 | ATC Level 4 | Preferred Name | Verbatim | Dose (Unit) | Route | Frequency | Given for AE or MH? |
| Reason for<br>Use | XXXXXXXX | | | | | | | | | | | | |
| Subject | XX-XXXX | | | | | | | | | | | | |
| Site | XXX | | | | | | | | | | | | |

ATC=Anatomical therapeutic class

Source: list SAS datasets used to create listing

DDMONYYYYTHH: MM

Program: program\_name

SAS X.Y

Programmer Note: AE and MH number should correspond to AESEQ and MHSEQ

Statistical Analysis Plan 402-C-413 (Page X of Y) Pacira Pharmaceuticals, Inc. EXPAREL Pacira Pharmaceuticals, Inc.  $EXPAREL^{\circledast}$ 

Listing 16.2-20.7: Concomitant Medications - All Subjects Cohort: cohort; Treatment: treatment-name

| | | Reason for | | |
|---|---|---|---|---|
| Site | Subject | Use | Data Type | Data |
| XXX | XX-XXX | XXXXXXXX | Start Date and Time | DDMONYYYYTHH:MM |
| | | | End Date and Time | DDMONYYYYTHH:MM |
| | | | Medication Number | × |
| | | | ATC Level 1 | XXXXXXXXXXXXXXXX |
| | | | ATC Level 2 | XXXXXXXXXXXXXXXXXX |
| | | | ATC Level 3 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | | ATC Level 4 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | | Preferred Name | XXXXXXXXXXXXXXXXXX |
| | | | Verbatim | XXXXXXXXXXXXXXXXXX |
| | | | Dose (Unit) | XXXXXXXX (XXXXXXXX) |
| | | | Route | XXXXXXXX |
| | | | Frequency | XXXXXXX |
| | | | Given for AE or MH? | XXXXXXXXXXXXXXX AE # XX (or MH # XX) |

ATC=Anatomical therapeutic class

Source: list SAS datasets used to create listing

DDMONYYYYTHH: MM

Program: program\_name

SAS X.Y

402-C-413 Statistical Analysis Plan Pacira Pharmaceuticals, Inc.  $\text{EXPAREL}^{\circledR}$ 

(Page X of Y) Pacira Pharmaceuticals, Inc. EXPAREL

402-C-413

Listing 16.2-21: Protocol Deviations - All Subjects Cohort: cohort; Treatment: treatment-name

| Description | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
|---------------|-----------------------------------------|
| Date and Time | DDMONYYYYHH:MM |
| Category | XXX |
| Subject | XX-YYYY |
| Site | XXX |

DDMONYYYYTHH: MM Program: program\_name Source: list SAS datasets used to create listing SAS X.Y

Note to programmer: Subjects may have multiple deviations. Sort deviations by cohort, treatment, center, subject.

| EXPAREL® | | Statistical Analysis Plan |
|---|---|---|
| Pacira Pharmaceuticals, Inc.<br>EXPAREL | (Page X of Y) | 402-C-413 |

Listing 16.2-22: Unique Adverse Events Terms and Associated Coded Terms

| MedDRA Terms | |
|---------------------------------|-----------------------------------------|
| SOC | |
| Preferred Term | Verbatim(s) |
| SOC1 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| PT1.1 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| PT1.2 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| SOC2 | |
| PT2.1 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| Coded using MedDRA version 22.0 | |

DDMONYYYYTHH: MM Program: program\_name Source: list SAS datasets used to create listing SAS X.Y

Note to programmer: Sort by SOC and preferred term in alphabetical order.

| 402-C-413 | Statistical Analysis Plan |
|---------------------------|---------------------------|
| Inc. | |
| Pacira Pharmaceuticals, I | EXPAREL® |

402-C-413 (Page X of Y) Pacira Pharmaceuticals, Inc. EXPAREL

Listing 16.2-23: Unique Medication Terms and Associated Coded Terms

Who Drug Dictionary Terms

ACT1

ACT2

ACT3

ACT4

Preferred name Verbatim(s)

ATC1.2 ATC1

PN1.2.1

ATC2

PN1.2.2

ATC2.2

ATC2.3

ATC2.4

PN2.2.3.4.1

Coded using Who Drug Dictionary Version March 2019 B3

Source: list SAS datasets used to create listing

DDMONYYYYTHH: MM

Program: program\_name

SAS X.Y

Note to programmer: Sort by ATC1, ATC2, ATC3, ATC4 and preferred name in alphabetical order

CONFIDENTIAL 68 of 68